CLINICAL TRIAL: NCT00490243
Title: A Randomized, Double-Blind Trial of the Effect of Different Anti-Asthmatic Treatments on Lung Function and on Exercise-Induced Bronchoconstriction in Children With Asthma
Brief Title: Effect of Different Anti-Asthmatic Treatments on Lung Function and on Exercise-Induced Bronchoconstriction in Children With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RNN/135/03/KE
Record Dates: First submitted 2007-06-21; First posted 2007-06-22 (Estimated); Last update posted 2007-06-28 (Estimated); Status verified 2007-06

CONDITIONS: Asthma
Keywords: Asthma; Children; Exercise; Pulmonary Function; Budesonide; Montelukast; Formoterol
MeSH Terms: conditions — Asthma; Motor Activity | interventions — Budesonide; montelukast; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: budesonide and montelukast
Drug: budesonide and formoterol
Drug: montelukast
Drug: budesonide
Drug: placebo

SUMMARY:
The present study was conducted to determine the effects of four week treatment with budesonide, montelukast, budesonide with montelukast and budesonide with formoterol in children with atopic asthma on lung function: forced expiratory volume in one second, mid-expiratory flow, peak expiratory flow rate, resistance by the interrupter technique, plethysmographic specific airway resistance, exercise-induced bronchial hyperreactivity and clinical symptoms.

DETAILED DESCRIPTION:
Asthma is one of the most common chronic disease worldwide, imposing a substantial social burden on children. Allergic inflammation is responsible for all clinical symptoms of asthma. The effects of allergic inflammation are: bronchial muscle constriction, excessive mucus production, and edema of mucosa, all elements of "asthmatic triad" causing bronchial obturation. Normal lung function is one of the goals of asthma management. In most of the studies the effect of monotherapy on the symptom scores, lung function parameters and bronchial hyperreactivity was assessed.

The present study was conducted to determine the effects of four week treatment with budesonide, montelukast, budesonide with montelukast and budesonide with formoterol in children with atopic asthma on lung function: forced expiratory volume in one second, mid-expiratory flow, peak expiratory flow rate, resistance by the interrupter technique, plethysmographic specific airway resistance, exercise-induced bronchial hyperreactivity and clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients
* Aged 6 to 18 with a clinical diagnosis of bronchial asthma with a duration of at least 6 months before the first visit and with current history of moderate persistent asthma
* Sensitive to house dust mites as shown by positive skin-prick tests to Dermatophagoides pteronyssinus or Dermatophagoides farinae
* To become eligible for the active treatment period, patients and their parents were required to do reproducible spirometry, whole body plethysmography and interrupter technique.
* In order to be included in the study the patients had to have a resting FEV1 of more or equal 70%.

Exclusion Criteria:

Study exclusions included:

* Active upper respiratory tract infection within 3 weeks before the study and acute sinus disease requiring antibiotic treatment within 1 month before the study
* Previous intubation
* Asthma hospitalisation during the 3 months before the first visit.
* Additional criteria were other clinically significant pulmonary, hematologic, hepatic, gastrointestinal, renal, endocrine, neurologic, cardiovascular, and/or psychiatric diseases or malignancy that either put the patient at risk when participating in the study or could influence the results of the study or the patient's ability to participate in the study as judged by the investigator.
* Excluded medications were β-blockers (eye drops included), astemizole within 3 months, or oral corticosteroids within 1 month before the first visit.
* Patients who were receiving immunotherapy were also excluded.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2003-07; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
FEF25-75%, Rint, sRaw, FEV1, PEFR, maximum percentage fall in FEV1 after exercise test, the area under the curve (AUC) for the FEV1 values over the 20-min period from exercise | baseline (second visit) and after 4 weeks of treatment (third visit)

SECONDARY OUTCOMES:
symptoms score | baseline (second visit) and after 4 weeks of treatment (third visit)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Grzelewski, MD, PhD, Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, Poland; Iwona Stelmach, MD, PhD, Prof, Study Chair — Department of Pediatrics and Allergy, Medical University of Lodz, Poland
Locations (1):
- Department of Pediatrics and Allergy, Medical University of Lodz, Poland, Lodz, Poland

REFERENCES:
- [Result] Stelmach I, Grzelewski T, Bobrowska-Korzeniowska M, Stelmach P, Kuna P. A randomized, double-blind trial of the effect of anti-asthma treatment on lung function in children with asthma. Pulm Pharmacol Ther. 2007;20(6):691-700. doi: 10.1016/j.pupt.2006.08.003. Epub 2006 Sep 14. PMID 17046300